CLINICAL TRIAL: NCT04888832
Title: Disparities in Medicaid and SNAP Participation: the Effects of Work Requirements and the COVID-19 Pandemic
Brief Title: The Effect of Work Requirements in SNAP in Virginia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: Abdul Latif Jameel Poverty Action Lab (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Tim Layton, 30th Anniversary Associate Professor of Health Care Policy, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB19-0859; 5R01MD014970-02 (NIH)
Record Dates: First submitted 2021-05-07; First posted 2021-05-17 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Health Disparities; Food Security
Keywords: Supplemental Nutrition Assistance Program; work requirements; Medicaid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Control Group (No Intervention): No change to work requirements or recertification period
- Intervention Group 1 (Active Comparator): Standard 6-month recertification period, additional 6-month work requirement exemption
  Interventions: Other: Work requirement exemption months
- Intervention Group 2 (Active Comparator): Standard 6-month recertification period, additional 12-month work requirement exemption
  Interventions: Other: Work requirement exemption months
- Intervention Group 3 (Active Comparator): Standard 6-month recertification period, additional 12-month work requirement exemption
  Interventions: Other: Work requirement exemption months
- Intervention Group 4 (Active Comparator): 12-month recertification period (6-month extension), additional 6-month work requirement exemption
  Interventions: Other: Work requirement exemption months

INTERVENTIONS:
Other: Work requirement exemption months — Cross-randomized intervention will test effect of additional exemption months before work requirements in SNAP become binding and extensions of the standard SNAP recertification period.
  Other Names: Change to recertification timeline
  Arms: Intervention Group 1; Intervention Group 2; Intervention Group 3; Intervention Group 4

SUMMARY:
More than a dozen states have proposed or plan to implement work requirements in Medicaid, and similar requirements already exist nationally in the Supplemental Nutritional Assistance Program (SNAP), yet evidence on the effects of these policies is limited. In cooperation with the state of Virginia, the investigators plan to conduct a randomized controlled trial studying the impacts of work requirements in public programs on insurance coverage, SNAP participation, employment, and health, with a particular focus on changes in racial/ethnic and geographic disparities in these outcomes. The COVID-19 epidemic and concurrent economic downturn creates additional urgency around these issues, and the investigators will use a combination of national administrative data and a new population survey to assess disparities in employment, health care, and food insecurity during this crisis.

DETAILED DESCRIPTION:
Work requirements are becoming increasingly common in major public assistance programs, with federal requirements for most adults to work in order to participate in the Supplemental Nutritional Assistance Program (SNAP, previously known as food stamps), and more than a dozen states proposing similar requirements in Medicaid. Proponents of work requirements contend that these policies increase beneficiary engagement in work and community activities that may lead to higher incomes and better health. On the other hand, opponents of work requirements suggest that many low-resource households will lose much-needed benefits, without commensurate improvements in employment. The investigators propose a randomized controlled trial of work requirements in Virginia, leveraging state support for exempting a portion of Medicaid expansion enrollees from the state's proposed work requirements. The investigators are also working with the state to explore the impact of work requirements in SNAP. They will study the impacts of each policy on health insurance coverage, access to care, employment, food insecurity, and health outcomes using a mix of administrative data and a new beneficiary survey. Our analysis will oversample several populations of interest, including racial/ethnic minorities and low-income rural residents. In doing so, investigators will identify the overall policy impacts of these policies, and will also assess who is most affected by each component to determine the impact of these policy changes on racial, ethnic, socioeconomic, and geographic disparities. Meanwhile, the COVID-19 epidemic and concurrent economic downturn create additional urgency around the issues of employment and participation in social programs. Using a combination of national administrative data and a new population survey, this study will also provide a timely assessment of disparities in employment, health care, and food insecurity during the current public health and economic crises.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for Virginia's SNAP program as an "able-bodied adult without dependents" (ABAWD) and thus subject to work requirements (this eligibility is age restricted to 18-49)

Exclusion Criteria:

* Categorical exemption from work requirements for any reason (e.g., has a disability, has dependents, resides in a geographic area where work requirements have been waived due to elevated employment)

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12500 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
SNAP enrollment | Up to 24 months after randomization
  Collected administratively (DSS records)
Employment status | Up to 24 months after randomization
  Collected administratively (VEC records)
UI covered earnings | Up to 24 months after randomization
  Collected administratively (VEC records)
Non-UI covered earnings | Up to 24 months after randomization
  Collected administratively (federal tax records)

SECONDARY OUTCOMES:
Number of jobs held | Up to 24 months after randomization
  Collected administratively (DSS records)
Medicaid participation | Up to 24 months after randomization
  Collected administratively (DSS records)
Hospitalizations | Up to 24 months after randomization
  Collected administratively (Virginia Health Information)
Credit scores | Up to 24 months after randomization
  Collected administratively (credit bureaus)
Evictions | Up to 24 months after randomization
  Collected administratively (court records)
Crime (records of charges, convictions) | Up to 24 months after randomization
  Collected administratively (court records)
Food insecurity | Survey to be administered approximately 1 year after randomization begins
  Collected by survey
Self-reported health | Survey to be administered approximately 1 year after randomization begins
  Collected by survey
Depression score | Survey to be administered approximately 1 year after randomization begins
  Collected by survey
Non-work community engagement activities | Survey to be administered approximately 1 year after randomization begins
  Collected by survey
Forced moves, housing instability | Survey to be administered approximately 1 year after randomization begins
  Collected by survey
Reasons for exiting SNAP | Survey to be administered approximately 1 year after randomization begins
  Collected by survey
Barriers to employment | Survey to be administered approximately 1 year after randomization begins
  Collected by survey
Hours worked per week | Survey to be administered approximately 1 year after randomization begins
  Collected by survey
Difficulty paying medical bills | Survey to be administered approximately 1 year after randomization begins
  Collected by survey
Uninsurance | Survey to be administered approximately 1 year after randomization begins
  Collected by survey

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Department of Social Services (Home Office), Glen Allen, Virginia, United States

IPD SHARING:
Plan to Share IPD: No